CLINICAL TRIAL: NCT01066364
Title: Colesevelam Versus Placebo in the Treatment of Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Rohit Loomba, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 091491
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: NASH; NAFLD; Steatohepatitis; Nonalcoholic; Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (sugar) pill (Placebo Comparator): Six tablets per day (identical to colesevelam)
  Interventions: Drug: Colesevelam Hcl
- Colesevelam arm (Experimental): 3.75 grams per day
  Interventions: Drug: Colesevelam Hcl

INTERVENTIONS:
Drug: Colesevelam Hcl — 3.75 gm/day (six 675 mg tablets)
  Other Names: Welchol

SUMMARY:
The purpose of the study is to see if the drug colesevelam is a potential treatment for Nonalcoholic Steatohepatitis(NASH).

DETAILED DESCRIPTION:
We plan to investigate the role of colesevelam, a bile-acid binding resin, in patients with NASH residing in the United States and assess liver fat changes during therapy using MRI of the liver. It can be hypothesized that colesevelam would lead to a greater improvement in insulin sensitivity and lipid profile compared with placebo and may lead to greater improvement in liver fat by MRI as compared to placebo.

In this pilot study, we propose to randomize approximately 55 patients (1:1 ratio) to either colesevelam or placebo and treat them for 24-weeks to evaluate changes in baseline insulin sensitivity, serum biochemistry (ALT and AST), and liver fat by MRI during therapy. Liver histologic changes would also be examined as an exploratory outcome for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age at entry at least 18 years.
2. Serum alanine (ALT) or aspartate (AST) aminotransferase activities that are above the upper limits of normal. 19 or more in women and 30 or more in men.
3. Evidence of hepatic steatosis or liver fat (>5%) by MRI.
4. Evidence of definite or suspected NASH
5. Written informed consent.

Exclusion criteria:

1. Evidence of another form of liver disease.
2. History of excess alcohol ingestion.
3. Contraindications to liver biopsy.
4. Decompensated liver disease.
5. History of gastrointestinal bypass surgery or ingestion of drugs known to produce hepatic steatosis.
6. Recent initiation or change of anti-diabetic drugs.
7. Use of colesevelam or other agents in the same class.
8. Significant systemic or major illnesses other than liver disease that, in the opinion of the investigator would preclude treatment with colesevelam and adequate follow up.
9. Positive test for anti-HIV.
10. Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year.
11. Pregnancy or inability to practice adequate contraception in women of childbearing potential.
12. Evidence of hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, MD, M.H.Sc, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - UCSD: Prevention Studies Clinic, La Jolla, California
  - UCSD: Medical Center- Hillcrest, San Diego, California

REFERENCES:
- [Derived] Nedrud MA, Chaudhry M, Middleton MS, Moylan CA, Lerebours R, Luo S, Farjat A, Guy C, Loomba R, Abdelmalek MF, Sirlin CB, Bashir MR. MRI Quantification of Placebo Effect in Nonalcoholic Steatohepatitis Clinical Trials. Radiology. 2023 Mar;306(3):e220743. doi: 10.1148/radiol.220743. Epub 2022 Nov 1. PMID 36318027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo (Sugar) Pill | Colesevelam Arm
Started | 25 | 25
Completed | 22 | 23
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Sugar) Pill | Colesevelam Arm | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.4) | 45.4 (12.7) | 47.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 11 | 19
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be Improvement in Hepatic Steatosis by Liver MRI
Description: To examine the efficacy of Colesevelam at 3.75 g/day orally versus placebo to decrease liver fat in patients with biopsy-proven nonalcoholic steatohepatitis.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: % of fat
Arm/Group | Placebo (Sugar) Pill | Colesevelam Arm
Number analyzed (Participants) | 22 | 24
% of fat | 17.9 (7.7) | 14.2 (6.3)

2. Secondary Outcome: Insulin Sensitivity as Determined by HOMA-IR
Description: To examine the efficacy of Colesevelam at 3.75 g/day orally versus placebo to decrease HOMA-IR in patients with biopsy-proven nonalcoholic steatohepatitis.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Sugar) Pill | Colesevelam Arm
Number analyzed (Participants) | 25 | 25
units on a scale | 8.3 (9.8) | 7.6 (12.3)

3. Secondary Outcome: Serum ALT and AST Values
Description: To examine the efficacy of Colesevelam at 3.75 g/day orally versus placebo to decrease serum ALT and AST in patients with biopsy-proven nonalcoholic steatohepatitis.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo (Sugar) Pill | Colesevelam Arm
Number analyzed (Participants) | 25 | 25
U/L
  ALT | 79.1 (47.8) | 86.6 (68.1)
  AST | 49.9 (32.1) | 56.2 (46.3)

4. Secondary Outcome: Lipid Profiles
Description: To examine the efficacy of Colesevelam at 3.75 g/day orally versus placebo to decrease improve the lipid profiles in patients with biopsy-proven nonalcoholic steatohepatitis.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Sugar) Pill | Colesevelam Arm
Number analyzed (Participants) | 25 | 25
mg/dL
  LDL | 115.8 (31.2) | 124.0 (37.7)
  Total Cholesterol | 202.4 (36.5) | 200.2 (46.0)

ADVERSE EVENTS:
Arm/Group | Placebo (Sugar) Pill | Colesevelam Arm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Sugar) Pill (N=25) | Colesevelam Arm (N=25)
Muscle ache with elevated CPK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Severe hot flashes with leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
IBD Exacerbation (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No